CLINICAL TRIAL: NCT07384936
Title: A Prospective, Controlled Study to Assess the Preliminary Efficacy and Safety of Topefilgrastim Injection in High-Risk Pregnant Patients With Preeclampsia.
Brief Title: Topefilgrastim Injection in the Treatment of High-Risk Pregnant Patients With Preeclampsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fang Wang (Other)
Collaborators: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Fang Wang, Chief physician, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG-5-1-005
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Topefilgrastim Injection
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Investigator-Initiated Trial (IIT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topefilgrastim 0.5mg Group (Experimental)
  Interventions: Drug: Topefilgrastim Injection
- Topefilgrastim 1mg Group (Experimental)
  Interventions: Drug: Topefilgrastim Injection
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Topefilgrastim Injection — Subjects will receive subcutaneous injection of 0.5 mg Topefilgrastim starting from Week 1 Day 1 (W1D1), with a frequency of once every two weeks, for at least 8 consecutive weeks.
  Arms: Topefilgrastim 0.5mg Group
Drug: Topefilgrastim Injection — Subjects will receive subcutaneous injection of 1 mg Topefilgrastim starting from Week 1 Day 1 (W1D1), with a frequency of once every two weeks, for at least 8 consecutive weeks.
  Arms: Topefilgrastim 1mg Group

SUMMARY:
This study is an open-label, prospective investigation designed to enroll 100 high-risk pregnant subjects with preeclampsia (PE). Participants will be allocated in a 2:2:1 ratio to one of three groups: the Topefilgrastim 0.5mg/biweekly group, the Topefilgrastim 1mg/biweekly group, or the control group, based on investigator judgment and patient preference. The overall study consists of three parts: a screening period, a treatment period, and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study, be able to understand, and sign the informed consent form.
* Aged 18 to 45 years (inclusive) at the time of signing the informed consent form.
* Assessed as high-risk for preeclampsia at gestational weeks 11-13, defined as either:

A risk value of ≥1/100 based on the simplified Fetal Medicine Foundation (FMF) model, OR A high-risk result from serum biomarker screening (sFlt-1, PLGF, sFlt-1/PLGF ratio). (See Appendix for details)

* Gestational weeks 11-13 at enrollment.
* Singleton intrauterine pregnancy (confirmed by transvaginal or transabdominal ultrasound).

Exclusion Criteria:

* History of psychiatric disorder not adequately controlled by medication.
* Unexplained vaginal bleeding at screening.
* Known uterine malformation.
* Evidence of positive serology for HIV, HBV (HBsAg positive), HCV (anti-HCV antibody positive), or syphilis.
* Known proliferative retinopathy.
* Presence of severe organic disease or any other condition that, in the judgment of the investigator, makes the subject unsuitable for study participation.
* Planned or current use of medications with potential drug-drug interactions with human granulocyte colony-stimulating factor (G-CSF) analogs, such as lithium.
* Known allergy to rhG-CSF products or their components, or allergy to recombinant human proteins/peptides derived from E. coli.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
soluble fms-like tyrosine kinase-1(sFlt-1) | Gestational weeks 11-13；15-17；24-28
placental growth factor(PLGF) | Gestational weeks 11-13；15-17；24-28
sFlt-1/PLGF ratio | Gestational weeks 11-13；15-17；24-28

SECONDARY OUTCOMES:
Incidence of preeclampsia | From 11 weeks of pregnancy to 6 weeks postpartum
Incidence of early-onset preeclampsia | From 11 weeks of pregnancy to 6 weeks postpartum
Incidence of PE-associated Preterm Delivery | From 11 weeks of pregnancy to 6 weeks postpartum
Miscarriage rate | From 11 weeks of pregnancy to 6 weeks postpartum
Preterm birth rate | From 11 weeks of pregnancy to 6 weeks postpartum
Gestational age at delivery | From 11 weeks of pregnancy to 6 weeks postpartum
Neonatal birth weight | From 11 weeks of pregnancy to 6 weeks postpartum
Incidence of small for gestational age (SGA) neonates | From 11 weeks of pregnancy to 6 weeks postpartum
Admission rate to the neonatal ward | From 11 weeks of pregnancy to 6 weeks postpartum
NICU admission rate | From 11 weeks of pregnancy to 6 weeks postpartum
Adverse Events (AEs) | From 11 weeks of pregnancy to 6 weeks postpartum
Serious Adverse Events (SAEs) | From 11 weeks of pregnancy to 6 weeks postpartum
Frequency of Adverse Events | From 11 weeks of pregnancy to 6 weeks postpartum
Frequency of Serious Adverse Events | From 11 weeks of pregnancy to 6 weeks postpartum
Severity of Adverse Events | From 11 weeks of pregnancy to 6 weeks postpartum
Severity of Serious Adverse Events | From 11 weeks of pregnancy to 6 weeks postpartum
Fetal Death | From 11 weeks of pregnancy to 6 weeks postpartum
Perinatal Death | From 11 weeks of pregnancy to 6 weeks postpartum
Incidence of congenital malformations | From 11 weeks of pregnancy to 6 weeks postpartum
Body Temperature | From 11 weeks of pregnancy to 6 weeks postpartum
Pulse | From 11 weeks of pregnancy to 6 weeks postpartum
Respiratory Rate | From 11 weeks of pregnancy to 6 weeks postpartum
Blood Pressure | From 11 weeks of pregnancy to 6 weeks postpartum
Height | From 11 weeks of pregnancy to 6 weeks postpartum
Weight | From 11 weeks of pregnancy to 6 weeks postpartum
Number of Participants with Abnormal Laboratory Parameters Findings | From 11 weeks of pregnancy to 6 weeks postpartum
Number of subjects with clinically significant abnormal findings in radiological examinations | From 11 weeks of pregnancy to 6 weeks postpartum
  including maternal/fetal or perinatal infants
Resistance Index (RI) of Uterine Spiral Arteries | Gestational weeks 11-13；15-17；24-28
Pulsatility Index (PI) of Uterine Arteries | Gestational weeks 11-13；15-17；24-28
Systolic to Diastolic Ratio (S/D ratio) of Uterine Spiral Arteries | Gestational weeks 11-13；15-17；24-28

CONTACTS AND LOCATIONS:
Overall Officials: Fang Wang, Principal Investigator — Lanzhou University Second Hospital
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, China